CLINICAL TRIAL: NCT01044797
Title: Remote Manipulation of a Capsule Endoscope in the Esophagus and Stomach of a Human Volunteer Using an External Hand-held Magnet
Brief Title: Remote Manipulation of a Capsule Endoscope
Acronym: Remote capsule
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Given Imaging (Unknown)
Responsible Party: Richard Rothstein, MD, Dartmouth-Hitchcock Medical Center
Other Study IDs: Given Imaging DHMC
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Healthy Volunteer; Given Capsule Manipulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to learn about the feasibility of moving a pill-sized camera (Givens Capsule) remotely in the esophagus and stomach using an external hand held magnet.

DETAILED DESCRIPTION:
Magnetic remote manipulation:

A simple and inexpensive method for manipulation of capsule endoscopes has been developed and successfully tested in survival studies in pigs. This has involved modifications of capsules which are in clinical use in patients as follows. One of the two imagers in esophageal capsules have been removed and replaced with three small magnets which are fixed within the capsule casing. This does not alter the dimensions of the capsule which can be reconstituted in a conventional casing. The magnetic reed switch which turns the capsule on and off is removed and is replaced with a thermal switch which will turn the capsule on if placed in hot water above 60 degrees centigrade for 60 seconds. The capsule can be manipulated using an external hand held paddle shaped magnet measuring approximately 20 x 20 x 5 centimeters which is held and rotated close to the back of the subject when the modified capsule is in the esophagus or the anterior abdominal wall when the capsule is in the stomach. The magnets used are of neodymium iron boron (quaternary ion magnets). The capsules are modified from FDA approved devices by Given Imaging (the company that makes these capsules). The outside of the capsule is unchanged but internal modifications, the changing of the switch and the inclusion of the magnet, are not FDA approved and are experimental.

Planned experiment in a human volunteer:

This study is for one, currently identified healthy volunteer only. The volunteer for this study is one of the inventors of the capsule endoscope technology (Paul Swain, MD) Dr. Swain will be consented in the usual manner with the current IRB approved consent. Dr. Rothstein will perform a physical exam to ensure that he is in general good health, has no esophageal or bowel disease or conditions that would contraindicate participation in the present study. He will then swallow a magnetically modified capsule as follows. He will be fasted overnight for the experiment which will be conducted in the designated endoscopy unit following standard endoscopic practise. A cannula will be placed for suitable intravenous access if needed, and D5/half normal saline infused to keep the vein open. The experiment will be performed with no sedation if possible or light sedation using benzodiazepines and/or narcotics (standard medications for endoscopy) at the discretion of the principal investigator and the volunteer. Topical anesthetics will be applied in the customary fashion for upper endoscopy. The volunteer will lie in the left lateral position and will swallow the capsule in a recumbent posture and may aid swallowing by sipping water from a glass through a straw. A flexible endoscope will be passed into the esophagus by the endoscopist. Another person who is not the endoscopist will manipulate the external paddle-shaped magnet. This involves moving and rotating the polarities of this magnet adjacent to the back and abdomen of the volunteer. A real-time viewer displaying images obtained from the capsule will be placed in a position so both the endoscopist and the paddle-magnet manipulator can view and react to the images. The images from the flexible endoscope, room images showing the movements of the paddle magnet and the real-time images acquired from the capsule will be recorded. The volunteer will be asked to indicate if he can feel the magnet moving the capsule in the esophagus and stomach and whether it is at all painful (real-time and via follow-up visual analog scale - pain 1 to10, 1 no pain and 10 worst pain).

The capsule will be manipulated in the esophagus and stomach with both flexible endoscopic and real time capsule imaging. Once manipulations in the esophagus have been completed the volunteer will be elevated (tilt table, sit or stand) to see if the magnet can hold the capsule in the esophagus against gravity. The capsule will then be allowed to pass into the stomach where it will be magnetically manipulated. Once the examination is completed the capsule will be removed using a Roth snare, a standardly employed accessory with a net which can be closed over objects for retrieval and is commonly used for polyp retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic adult volunteer with previously determined normal esophagus and stomach who understands the risks of the procedure.

Exclusion Criteria:

* Known strictures in the intestine,
* Crohn's disease,
* Swallowing difficulty,
* Age less than 21,
* Age over 75 or have a pacemaker,
* Presence of implanted metal devices,
* Presence of esophageal or bowel disease or conditions that may preclude study participation as a matter of clinical judgment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: One Human Volunteer, Healthy
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard I Rothstein, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center